CLINICAL TRIAL: NCT05235997
Title: A Multiple-Dose, Randomized, Double-Blinded, Placebo Controlled Trial To Evaluate The Efficacy Of Hydrolyzed Collagen Peptide In Adult Females
Brief Title: Placebo Controlled Efficacy Evaluation of the Hydrolyzed Collagen Peptide In Adult Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sel Sanayi Urunleri Ticaret ve Pazarlama A.S. (Industry)
Collaborators: Alpan Farma Ar-Ge Biyoteknolojileri Ltd.Sti. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ALP-2021-CL-01-2021/01997
Record Dates: First submitted 2022-01-07; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Skin; Skin Manifestations; Wrinkle
MeSH Terms: conditions — Skin Manifestations | interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolized Collagen Peptide (Experimental): This arm will be allocated randomly and receive 10 g hydrolized collagen peptide (Investigational Product) daily throughout the study.
  Interventions: Dietary Supplement: Hydrolized Collagen Peptide
- Placebo (Placebo Comparator): This arm will be allocated randomly and receive placebo throughout the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolized Collagen Peptide — Dietary Hydrolized Collagen Peptide sourced from bovine
  Other Names: Collagen
  Arms: Hydrolized Collagen Peptide
Other: Placebo — Placebo look alike the experimental product
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the contribution of hydrolized collagen products to elasticity, hydration and roughness of the skin of female volunteers. Safety and tolerability of the product is the other objective of this placebo-controlled, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers aged between 35 and 60 years,
* Volunteers who have normal physical examination at screening visit,
* Volunteers who have ability to communicate adequately with the investigator and in agreement to comply with the study requirements,
* Volunteers who have normal blood pressure and heart rate measured under stabilised conditions at the screening visit after at least 5 minutes of rest under supine position: SBP within 100 to 140 mmHg, DBP within 60 to 90 mmHg and HR within 50 to 100 bpm at least after 5 minutes of rest,
* Volunteers who have understanding of the study and agreement to give a written informed consent.

Exclusion Criteria:

* Who have atopic constitution or asthma and/or known allergy for biosynthetic collagen products and/or other any of the excipients of the product.
* Who have hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Who have the use of oral retinoids or oral steroids in the 6 months prior to initiation of the study.
* Who have the use of topical retinoids, anti-wrinkle cosmetic products including retinol and/or AHA, or moisture-rich cosmetic products within the 3 months prior to initiation of the study.
* Who use skincare therapy using lasers or peeling within the 3 months prior to initiation of the study.
* Who have current participation in another clinical study, or participation in any type of dermatology study within 3 months.
* Who have any history or presence of clinical relevance of cardiovascular, neurological, musculoskeletal, haematological, hepatic, gastrointestinal, renal, pulmonary, endocrinological, metabolism or psychiatric disease, any type of porphiria.
* Who have the presence or history of malabsorption or any gastrointestinal surgery except appendectomy or except herniotomy.
* Who had undergone, or planned to undergo, pregnancy or breastfeeding.
* Who have current intake of contraceptives, female hormones, obesity drugs, absorption inhibitors, antidepressants, or appetite suppressants.
* Who are suspected to have a high probability of non-compliance to the study procedure and/or completion of the study according to the investigator's judgment.
* Who have history of drug abuse.
* Who have relationship to the investigator.
* Who are not suitable to any of inclusion criteria.
* Who have history of difficulty of swallowing.
* Who are on a special diet due to any reason, or, have gained or lost 5% of baseline weight.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change on skin elasticity | 3 months
  Measurement of elasticity based on the stress/deformation method through skin suction by using an instrument specifically developed for assign skin health.
Change on skin hydration | 3 months
  Measurement is based on the hydration of the stratum corneum through the capacitive method by using an instrument specifically developed for assign skin health.

SECONDARY OUTCOMES:
Change on skin roughness | 3 monhs
  Measurement is based on capturing skin images by using an instrument specifically developed for assign skin health.

OTHER OUTCOMES:
Adverse events | 3 months
  Safety and tolerability of Hydrolized Collagen Peptide

CONTACTS AND LOCATIONS:
Locations (1):
- Huseyin Serhat Inaloz, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No